CLINICAL TRIAL: NCT06384287
Title: Effects of Therapeutic Hemodynamic Interventions on Peripheral Perfusion in Intensive Care
Brief Title: Peripheral Tissue Perfusion in Intensive Care
Acronym: INPPEREA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231342
Record Dates: First submitted 2024-04-03; First posted 2024-04-25 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Circulatory Failure
Keywords: Tissue perfusion; Capillary refill time; Skin blood flow; Fluid challenge; Inotrope
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Fluid challenge: Impact of fluid challenge on peripheral tissue perfusion on sepsis patients
- Vasopressors: Impact of vasopressors on peripheral tissue perfusion on sepsis patients
- Inotrope: Impact of dobutamine on peripheral tissue perfusion on patients with septic or cardiogenic shock

SUMMARY:
Tissue perfusion has been identified as an early prognosis factor in patients admitted to intensive care. However, little is known about the effects of different hemodynamic interventions performed in clinical routine on peripheral tissue perfusion.

The aim of this work is to study the kinetics of CRT and local skin blood flow following therapeutic intervention (fluid challenge, vasopressor or inotropic drug).

DETAILED DESCRIPTION:
Sepsis is today a major cause of morbidity and mortality worldwide. Septic shock, the most serious manifestation of the infection, affects 2 to 20% of intensive care patients. Despite appropriate antibiotic therapy and improved resuscitation strategies based on early treatment, volume expansion and rational use of vasopressors, the mortality rate of shock states remains too high, between 40 and 50%.

Over the past two decades, great advances have been made in the understanding the pathophysiology of septic shock. Microcirculatory abnormalities have been identified as the main cause of organ hypoperfusion and visceral failure leading to death. In addition, several studies in animals and humans have highlighted a discordance between systemic hemodynamic parameters and alterations of small vessels during shock suggesting that microvascular blood flow and tissue perfusion should be analyzed in patients with acute circulatory failure in association with blood pressure and cardiac output. Capillary refill time (CRT), is an easy-to-use, easy-to learn tool to evaluate peripheral tissue perfusion. CRT is a strong predictive factor of organ failure severity and poor outcome in critically ill patients with sepsis. A recent randomized trial reported promising results regarding the use of CRT to guide resuscitation. However, little is known about the impact of treatment on CRT. The aim of this work is to study the kinetics of CRT and local skin blood flow following therapeutic intervention (fluid challenge, vasopressor or inotropic drug).

ELIGIBILITY:
Inclusion Criteria:

* Patients in intensive care unit with acute circulatory failure related to sepsis or cardiac failure requiring therapeutic intervention

Exclusion Criteria:

* Agitation
* Hemorrhagic shock
* Severe skin lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care unit with acute circulatory failure related to sepsis or cardiac failure requiring a therapeutic intervention (fluid challenge or vasopressor or dobutamine)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Skin blood flow variations | continuous monitoring during 1 hour maximum starting just before intervention
  Measurement using laser doppler probe in the finger tip

SECONDARY OUTCOMES:
Capillary refill time | at baseline, 3 timepoints after starting interventions (10, 30 and 60 minutes)
  Clinical measurement at bedside
Mottling score | at baseline, 3 timepoints after starting interventions (10, 30 and 60 minutes)
  Clinical measurement at bedside
correlation between Skin blood flow and CRT (baseline and variations) | at baseline, at 10, 30 and 60 minutes after intervention
  Measurement using laser doppler probe in the finger tip
correlation between skin blood flow and Cardiac output | at baseline, at 10, 30 and 60 minutes after intervention
  Laser doppler with skin probe and echocardiography
correlation between skin blood flow and mean arterial pressure | at baseline, at 10, 30 and 60 minutes after intervention
  Laser doppler with skin probe and arterial catheter

CONTACTS AND LOCATIONS:
Locations (1):
- Saint -Antoine Hospital_Médecine Intensive Reanimation, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided